CLINICAL TRIAL: NCT00674219
Title: Differential Efficacy of Memantine for Obsessive-compulsive Disorder vs. Generalized Anxiety Disorder: an Open-label Trial
Brief Title: Memantine Treatment for Obsessive-compulsive Disorder and Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Saban Family Foundation (Other)
Responsible Party: Principal Investigator, Alexander Bystritsky, Professor of Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-08-063-03
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Obsessive-Compulsive Disorder; Generalized Anxiety Disorder
Keywords: Obsessive-compulsive disorder; Generalized anxiety disorder; Memantine; Namenda
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Generalized Anxiety Disorder | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCD group (Active Comparator): OCD group - received 12 weeks of open-label memantine 10 mg twice daily, as either mono therapy or augmentation of their existing medication.
  Interventions: Drug: Memantine
- GAD group (Active Comparator): GAD group - received 12 weeks of open-label memantine 10 mg twice daily, as either mono therapy or augmentation of their existing medication.
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Namenda 10mg BID for 12 weeks
  Other Names: Namenda

SUMMARY:
The objective of this study was to obtain preliminary open-label data on the efficacy and tolerability of memantine, an anti-glutamatergic medication with a unique pharmacodynamic profile, in individuals with OCD and individuals with GAD. Because glutamatergic hyperactivity in frontal and frontal-subcortical circuits may play a role in the symptomatic expression of OCD, and possibly GAD, agents that reduce glutamatergic neurotransmission should provide unique anti-stress and anti-obsessional benefits. Memantine is a specific, uncompetitive antagonist at the NMDA receptor that blocks sustained activation of the NMDA receptor by high concentrations of glutamate under pathological conditions but rapidly leaves the NMDA channel upon transient physiological activation by low concentrations of glutamate.

DETAILED DESCRIPTION:
Several case reports and an open-label trial have reported efficacy of anti-glutamatergic medications for the treatment of OCD. In an open-label trial of riluzole, a glutamate release inhibitor, seven of 13 adult patients with OCD improved, and five were categorized as treatment responders. Another open trial found riluzole to be effective for four of six children with treatment-refractory OCD. N-acetylcysteine, an agent that likely attenuates glutamate neurotransmission, was effective as an augmentation in one patient with OCD. Two case reports described memantine treatment of OCD. Poyurovsky et al. reported improvement with memantine augmentation in one patient with treatment resistant OCD, while Pasquini and Biondi noted improvement in one OCD patient with checking compulsions but not in one with contamination obsessions. There have been no controlled or open-label trials of memantine in OCD reported thus far.

Few studies have examined the efficacy of anti-glutamatergic agents in GAD. In an open-label trial of riluzole treatment in 18 patients with GAD, twelve patients responded and eight achieved remission. A double-blind, controlled study found that LY354740, a metabotropic glutamate receptor 2/3 (mGlu2/3) agonist, was significantly more effective than placebo for GAD. No studies of memantine in GAD have been reported thus far. We hypothesized that treatment with memantine would result in significant symptom reduction in both OCD and GAD.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female outpatient between 18-64 years old.
* The subject meets DSM-IV criteria for Generalized Anxiety Disorder or Obsessive Compulsive Disorder as determined by the MINI.
* Sexually active female patients of childbearing potential must be practicing at least one or more the following methods of contraception during the study: intrauterine device (IUD), barrier method in combination with a spermicide, oral/hormonal contraception or abstinence. Female patients of childbearing potential must have a negative pregnancy test prior to receiving study drug.
* Written informed consent must be obtained from the subject prior to study participation.
* The subject is in good medical health or with chronic medical conditions which are currently stable.
* No current abuse of alcohol or other substance.
* The subject has a total score of 20 or more on the HARS or YBOCS at screening (for GAD and OCD, respectively)
* The subject has a Clinical Global Impression (CGI) Severity score of 4 or more at screening.

Exclusion Criteria:

* The subject meets DSM-IV criteria for an Axis I diagnosis (other than GAD or OCD) as the primary diagnosis (i.e., schizophrenia, mood disorder, psychosis, anorexia nervosa) as determined by the MINI.
* The subject is clinically judged by the investigator to be at risk for suicide or is acutely suicidal as objectively measured by the MINI and MSE.
* The subject is clinically judged by the investigator to be at risk for homicide or is acutely homicidal as objectively measured by the MINI and MSE.
* The subject has a psychiatric condition that would require inpatient, or partial psychiatric hospitalization.
* Seizure disorders.
* Significant history of medical disease (i.e. cardiovascular, hepatic (e.g. cirrhosis, hepatitis B or C) renal, gynecological, musculoskeletal, neurological, gastrointestinal, metabolic, hematological, endocrine, cancer with a metastatic potential or progressive neurological disorders) which could impair reliable participation in the trial or necessitate the use of medication not allowed by this protocol.
* The subject is pregnant, planning to become pregnant, or nursing. If a subject becomes pregnant, she will be discontinued immediately and followed appropriately.
* Concomitant therapy with another investigational drug, or participation in an investigational drug study within one month prior to entering this study.
* Current psychotherapeutic treatment except for treatment with Specific Reuptake Inhibitor (SSRIs) medications which include: Fluoxetine (Prozac), Paroxetine (Paxil), Sertraline (Zoloft), Luvox (Fluvoxamine), and Citalopram. Potential subjects may remain on one of the SSRI medications provided that he or she has been on a stable dose for at least 4 weeks prior to entering this study; this dose remains stable throughout the remainder of this study; and it can be determined that this medication is not exacerbating the anxiety symptoms.
* History of poor compliance or in the Investigator's judgment patients any subject whose treatment as an outpatient would be clinically contraindicated
* The subject has attempted suicide one or more times within the past twelve months
* The subject has a Structured Hamilton Depression Rating Scale (SIGH-D) score above 38 which suggests a moderate to severe clinical level of depressive symptoms

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bystritsky, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feusner JD, Kerwin L, Saxena S, Bystritsky A. Differential efficacy of memantine for obsessive-compulsive disorder vs. generalized anxiety disorder: an open-label trial. Psychopharmacol Bull. 2009;42(1):81-93. PMID 19204653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited during 2007-2008 from the Anxiety Disorders Program at UCLA.
Groups:
- OCD Group: Persons meeting inclusion criteria for a diagnosis of obsessive-compulsive disorder.
- GAD Group: Persons meeting inclusion criteria for a diagnosis of generalized anxiety disorder.
Period: Overall Study
Arm/Group | OCD Group | GAD Group
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Persons meeting inclusion criteria for a diagnosis of OCD or GAD.
Groups:
- Total: Total of all reporting groups
Arm/Group | OCD Group | GAD Group | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Mean (Full Range); unit: years] — Age of participants was collected but was not a predictor of study outcomes.
  years | 38.6 [18 to 64] | 37 [18 to 64] | 37.9 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of participants was collected but was not a predictor of study outcomes.
  Participants
    Female | 6 | 5 | 11
    Male | 4 | 2 | 6
Diagnosis of OCD or GAD [Number; unit: participants] — The Yale-Brown Obsessive Compulsive Scale (YBOCS) for the OCD group; the Hamilton Anxiety Rating Scale (HARS) for the GAD group; and the Clinical Global Impression-Improvement Scale (CGII) for both groups
  participants | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Psychometric Scores
Description: Participants in the OCD group were rated using the Yale-Brown Obsessive Compulsive Scale (Y-BOCS), a standard measure of obsessive-compulsive disorder (OCD) severity in pharmacotherapy studies. It is administered by a trained rater. It comprises 10 items assessing OCD symptoms (e.g. time spent, degree of control, severity). Each item is scored on a scale from 0 (not present) to 4 (severe) [total score range = 0-40] over the previous week. The higher the number on the Y-BOCS, the more severe the symptoms.
  Participants in the GAD group were rated using the Hamilton Anxiety Rating Scale (HARS), a standard measure of anxiety severity in pharmacotherapy studies. It is administered by a trained rater. It comprises 14 items assessing anxiety symptoms. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- OCD Group: Persons meeting inclusion criteria for a diagnosis of OCD.
- GAD Group: Persons meeting inclusion criteria for a diagnosis of GAD.
Arm/Group | OCD Group | GAD Group
Number analyzed (Participants) | 10 | 7
units on a scale
  12 weeks | 16.4 (13.6) | 18.86 (4.14)
  Baseline | 27.6 (4.4) | 24.3 (1.7)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | OCD Group | GAD Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 3/10 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCD Group (N=10) | GAD Group (N=7)
dizziness (Nervous system disorders) | 3 (3) | 3 (3)
Somnolence (Nervous system disorders) | 2 (3) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes